CLINICAL TRIAL: NCT03617588
Title: A Phase II, Open-label Study to Assess Safety and Clinical Utility of 68Ga-THP-PSMA PET/CT in Patients With High Risk Primary Prostate Cancer or Biochemical Recurrence After Radical Treatment (PRONOUNCED Study)
Brief Title: 68Ga-THP-PSMA PET/CT Imaging in High Risk Primary Prostate Cancer or Biochemical Recurrence of Prostate Cancer
Acronym: PRONOUNCED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theragnostics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: THERAG0001
Record Dates: First submitted 2018-06-21; First posted 2018-08-06 (Actual); Results first posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gallium-68 THP-PSMA (Experimental): Single intravenous administration of Gallium-68 THP-PSMA
  Interventions: Drug: Gallium-68 THP-PSMA

INTERVENTIONS:
Drug: Gallium-68 THP-PSMA — Subjects will undergo a Gallium-68 THP-PSMA scan in addition to standard of care monitoring. The results of this scan may influence the patient management plan.
  Other Names: THG-001

SUMMARY:
This will be an open-labelled, single centre study in the UK. The study group will include 60 patients with three groups of patients being studied. Group A will consist of 20 patients who have been newly diagnosed with primary high risk prostate cancer and are scheduled for radical prostatectomy surgery. Group B will consist of 20 patients with a diagnosis of BCR with previous radical prostatectomy, and are being considered for radical salvage therapy. Group C will consist of 20 patients with a diagnosis of BCR with previous radical radiotherapy (but no surgery), and are being considered for radical salvage therapy.

ELIGIBILITY:
Inclusion Criteria:

Group A: Adenocarcinoma of the prostate gland suitable for radical Tx.

* Adenocarcinoma of Prostate
* Gleason score 4+3 and above, or PSA > 20 ng/mL or clinical stage >T2C.
* Suitable for surgical tx
* No Hormone Therapy in last 3 months

Group B: PCa and a diagnosis of BCR, previously treated with radical prostatectomy, being considered for radical salvage therapy (with curative intent).

* Original diagnosis of PCa, treated with radical curative therapy at least 3 months before enrolment, and has been diagnosed with BCR based on:

  1. Post RP: two consecutive rises in PSA and final PSA >0.lng/ml OR Post RP: three consecutive rises in PSA. This definition is also applicable to subjects with PSA persistence post RP (where the PSA fails to fall to undetectable levels).
  2. Post RP: PSA doubling time of ~15 months OR PSA level 0.5 ng/ml.
* No previous recurrences of PCa.
* Consideration for radical salvage therapy.
* Should not have received androgen-deprivation therapy within 3 months of screening.
* No Hormone Therapy in last 3 months

Group C: PCa and a diagnosis of BCR, previously treated with radical radiotherapy, being considered for radical salvage therapy (with curative intent).

* The subject has had an original diagnosis of PCa and underwent radical curative therapy at least 3 months before enrolment, and has been diagnosed with BCR on the basis of:
* Increase in PSA level ~2.0 ng/ml above the nadir level after radiotherapy (RT) or brachytherapy, no previous recurrences of BCR.
* The subject is being considered for radical salvage therapy.
* Should not have received androgen-deprivation therapy within 3 months of screening.
* No hormone therapy within the past three months.

Exclusion Criteria:

Group A:

* Prior Tx for Prostate Tumours
* Gleason < 4+3
* Hip prostheses
* eGFR <20

Group B:

* Hormone Therapy in the last 3 months
* Hip prostheses
* eGFR <20

Group C:

* Hormone Therapy in the last 3 months
* Hip prostheses
* eGFR <20

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 49 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - St Bartholomew's Hospital (PIC), London
  - Royal Free Hospital (PIC), London
  - Guy's and St Thomas' Hospital (PIC), London
  - University College Hospital London, London

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period June 18th 2018 to June 12th 2019.
Groups:
- Group A: Patients with newly diagnosed primary high-risk PCa who were scheduled for RP surgery.
- Groups B and C: Group B: Patients with PCa and a diagnosis of BCR, previously treated with RP and being considered for radical salvage therapy (with curative intent).
  Group C: Patients with PCa and a diagnosis of BCR, previously treated with radical radiotherapy and being considered for radical salvage therapy (with curative intent).
Period: Overall Study
Arm/Group | Group A | Groups B and C
Started | 20 | 29
Completed | 19 | 29
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Groups B and C | Total
Number analyzed (Participants) | 20 | 29 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 14 | 22
  >=65 years | 12 | 15 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 29 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 13 | 21 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 29 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Management
Description: The impact of 68Ga-THP-PSMA PET/CT on the management of patients with PCa was analysed by measuring the percentage of patients who had a change in management plan as a result of 68Ga-THP-PSMA PET/CT documented after scan, compared with their pre-scan management plan. A change status of 'Yes' was assigned if there was any difference in treatment options between the intended and revised management plans. A change status of 'No' was assigned if the intended and revised management plans remained identical. This endpoint was assessed in the full analysis set, but as a sensitivity analysis, was also assessed in the per protocol population in case there was a difference between the populations. As all 49 patients underwent a technically successful post-baseline scan, the full analysis set and per protocol populations were the same.
Time Frame: up to 3 months post PET/CT
Population: Subject analysis set title:
  Safety Evaluable Population
  Subject analysis set type:
  Safety analysis
  Subject analysis set description:
  All patients who received a 68Ga-THP-PSMA PET/CT dose, regardless of whether they received the full intended dose, or proceeded to undergo the intended 68Ga-THP-PSMA PET/CT scan.
Measure: Count of Participants; unit: Participants
Groups:
- Full Analysis Set: A subset of the safety population who underwent the Visit 2 68Ga-THP-PSMA PET/CT scan, regardless of whether the scan was a technical success or failure.
- Per Protocol Set: A subset of the Full Analysis Set with at least one technically successful post baseline 68Ga-THP-PSMA PET/CT scan and without any major protocol deviations.
Arm/Group | Group A | Groups B and C | Full Analysis Set | Per Protocol Set
Number analyzed (Participants) | 20 | 29 | 49 | 49
Participants
  change in management plan | 6 | 15 | 21 | 21
  no change in management plan | 14 | 14 | 28 | 28

2. Secondary Outcome: Safety - Treatment Emergent Adverse Events
Description: Safety was assessed by means of physical examination, vital signs, cardiovascular profile, performance status, laboratory evaluations (haematology, biochemistry, urinalysis and prostate-specific antigen), recording of concurrent illness/therapy and AEs. No dose limiting toxicity was defined in this study.
Time Frame: Safety was assessed at screening, during the study and at Visit 4. AEs, regardless of relationship to study treatment, were recorded from the time of 68Ga-THP-PSMA administration until 30 days after the administration of 68Ga-THP-PSMA.
Measure: Number; unit: number of subjects
Groups:
- Safety Evaluable Population: All patients who received a 68Ga-THP-PSMA PET/CT dose, regardless of whether they received the full intended dose, or proceeded to undergo the intended 68Ga-THP-PSMA PET/CT scan.
Arm/Group | Group A | Groups B and C | Safety Evaluable Population
Number analyzed (Participants) | 20 | 29 | 49
number of subjects
  Any TEAE | 2 | 3 | 5
  Any TEAE related to 68Ga-THP-PSMA | 1 | 1 | 2
  Any TEAE CTCAE Grade 3 or higher | 1 | 1 | 2
  Any related TEAE CTCAE Grade 3 or higher | 0 | 0 | 0
  Any TEAE with outcome of death | 0 | 0 | 0
  Any related TEAE with outcome of death | 0 | 0 | 0
  Any serious TEAE | 0 | 0 | 0
  Any serious TEAE related to 68Ga-THP-PSMA | 0 | 0 | 0
  Any TEAE leading to discontinuation from study | 0 | 0 | 0
  Any related TEAE leading to discontinuation | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Safety was assessed at screening, during the study and at Visit 4. AEs, regardless of relationship to study treatment, were recorded from the time of 68Ga-THP-PSMA administration until 30 days after the administration of 68Ga-THP-PSMA.
Description: Safety was assessed by means of physical examination, vital signs, cardiovascular profile, performance status, laboratory evaluations (haematology, biochemistry, urinalysis and prostate-specific antigen), recording of concurrent illness/therapy and AEs. No dose limiting toxicity was defined in this study.
Arm/Group | Group A | Groups B and C | Safety Evaluable Population
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/29 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/29 | 0/49
Other Adverse Events (participants affected / at risk) | 2/20 | 3/29 | 5/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=20) | Groups B and C (N=29) | Safety Evaluable Population (N=49)
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Sensory loss (Nervous system disorders) | 0 | 1 | 1
Catheter site rash (General disorders) | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT03617588/SAP_000.pdf
  • Study Protocol (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT03617588/Prot_001.pdf